CLINICAL TRIAL: NCT07120763
Title: Pain Control Alternatives in Pediatric Patients With Distal Radius Fractures
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Tara Petroski, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00009073
Record Dates: First submitted 2025-04-15; First posted 2025-08-13 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Distal Radius Fracture Reduction; Pain Control; Pediatric Fractures
MeSH Terms: conditions — Agnosia | interventions — Ketamine; Lidocaine; Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Full ketamine sedation (Active Comparator): Including group of patients treated with full ketamine sedation in setting of distal radius fracture reduction
  Interventions: Drug: Ketamine group
- Hematoma block/minimal ketamine pain control (Active Comparator): Including group of patients treated with hematoma block/minimal ketamine pain control (. 0.25mg/kg) for distal radius fracture reduction in pediatric patients requiring reduction
  Interventions: Drug: Ketamine + Lidocaine
- hematoma block/intranasal fentanyl (Active Comparator): Including control group of patients treated with intranasal fentanyl and hematoma block, utilized in the setting of distal radius fractures in pediatric patients requiring reduction
  Interventions: Drug: Fentanyl (Nasalfent, Fentanyl Citrate Nasal Spray)

INTERVENTIONS:
Drug: Ketamine + Lidocaine — Including comparisons between patients randomized for treatment with full ketamine sedation in setting of distal radius fracture reduction, hematoma block/minimal ketamine pain control (. 0.25mg/kg) for distal radius fracture reduction, or intranasal fentanyl and hematoma block, utilized in the setting of distal radius fractures in pediatric patients requiring reduction
  Arms: Hematoma block/minimal ketamine pain control
Drug: Ketamine group — Including comparisons between patients randomized for treatment with full ketamine sedation in setting of distal radius fracture reduction, hematoma block/minimal ketamine pain control (. 0.25mg/kg) for distal radius fracture reduction, or intranasal fentanyl and hematoma block, utilized in the setting of distal radius fractures in pediatric patients requiring reduction
  Arms: Full ketamine sedation
Drug: Fentanyl (Nasalfent, Fentanyl Citrate Nasal Spray) — Including comparisons between patients randomized for treatment with full ketamine sedation in setting of distal radius fracture reduction, hematoma block/minimal ketamine pain control (. 0.25mg/kg) for distal radius fracture reduction, or intranasal fentanyl and hematoma block, utilized in the setting of distal radius fractures in pediatric patients requiring reduction
  Other Names: fentanyl + lidocaine
  Arms: hematoma block/intranasal fentanyl

SUMMARY:
The aim of this study is to evaluate the efficacy of a hematoma block and minimal ketamine pain control or hematoma block and intranasal fentanyl in pediatric patients presenting with distal radius fractures requiring reduction, compared to control of standard full conscious sedation using ketamine.

ELIGIBILITY:
Inclusion Criteria:

* Children requiring reduction for distal radius fracture
* Children presenting to the emergency department
* Children who are ages 3 to 17 years.

Exclusion Criteria:

* Pediatric patients <3 years old
* Adult patients (i.e. ages 18 or up)
* Pediatric patients with injury patterns that are not amenable to hematoma block.
* Children who are not a candidate for sedation related to BMI > 95%tile for age, ASA class > 2, Mallampati score > 2, and pregnant patients

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-08-22 (Actual); Primary Completion 2026-08-22 (Estimated); Study Completion 2027-08-22 (Estimated)

PRIMARY OUTCOMES:
Pain control efficacy | 1 hour after fracture reduction is complete on the day of the procedure/study visit.
  Including control group of patients treated with full ketamine sedation in setting of distal radius fracture reduction; randomization of patients deemed safe for full sedation to either control group, or one of two intervention groups including (group 1) hematoma block/minimal ketamine pain control (0.25mg/kg), and (group 2) intranasal fentanyl and hematoma block, utilized in the setting of distal radius fractures in pediatric patients requiring reduction. The investigators will be obtaining Visual Analog Scale (VAS) pain scores for each group to determine pain control efficacy and to compare between groups. This is a numeric pain scale with associated faces to help children determine their pain level, with 0 being "no pain" (with a smiley/happy face) and 10 being "most pain possible" (with a sad/crying face).
Patient satisfaction scores | 1 hour after fracture reduction is complete on the day of the procedure/study visit.
  Including control group of patients treated with full ketamine sedation in setting of distal radius fracture reduction; randomization of patients deemed safe for full sedation to either control group, or one of two intervention groups including (group 1) hematoma block/minimal ketamine pain control (0.25mg/kg), and (group 2) intranasal fentanyl and hematoma block, utilized in the setting of distal radius fractures in pediatric patients requiring reduction. The investigators will be obtaining patient satisfaction scores via a 5-point Likert scale to compare patient satisfaction between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Oshei Children's Hospital, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared. This is a single institution study; results will be shared after de-identification/analysis in the form of publication/presentation.

REFERENCES:
- [Background] McCarty EC, Mencio GA, Walker LA, Green NE. Ketamine sedation for the reduction of children's fractures in the emergency department. J Bone Joint Surg Am. 2000 Jul;82-A(7):912-8. doi: 10.2106/00004623-200007000-00002. PMID 10901305
- [Background] Disel NR, Yilmaz HL, Sertdemir Y, Yesilagac H, Avci A. Etomidate Versus Ketamine: Effective Use in Emergency Procedural Sedation for Pediatric Orthopedic Injuries. Pediatr Emerg Care. 2016 Dec;32(12):830-834. doi: 10.1097/PEC.0000000000000373. PMID 25834964
- [Background] Jordan RW, Aquilina A, Westacott DJ, Cooke S. A comparison of ketamine sedation and general anaesthesia for manipulation of paediatric forearm fractures. Acta Orthop Belg. 2016 Dec;82(4):836-842. PMID 29182126
- [Background] Morrison T, Carender C, Kilbane B, Liu RW. Procedural Sedation With Ketamine Versus Propofol for Closed Reduction of Pediatric Both Bone Forearm Fractures. Orthopedics. 2017 Sep 1;40(5):288-294. doi: 10.3928/01477447-20170824-01. Epub 2017 Sep 7. PMID 28877328
- [Background] Kwong A, Aldridge ES, Jayawardana R, Brookwick A, Miller J, Buntine PG. Length of stay outcomes in patients receiving ketamine sedation versus Bier's block anaesthesia for procedural closed fracture reduction: A retrospective audit of paediatric emergency department patients. Emerg Med Australas. 2022 Feb;34(1):73-77. doi: 10.1111/1742-6723.13844. Epub 2021 Aug 29. PMID 34459117